CLINICAL TRIAL: NCT01927484
Title: Methotrexate in Hand Osteoarthritis
Brief Title: Hand OA AND Methotrexate Use
Acronym: Hand OA & MTX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID-19 Pandemic
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, MD, University of Alexandria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: alexmed1391963211975
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Reduction in Pain; Reduction of Inflammation; Improvement in Function
Keywords: methotrexate,; osteoarthritis,; pain,; function,; synovitis
MeSH Terms: conditions — Osteoarthritis; Pain; Synovitis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methotrexate (Experimental): 25mg oral methotrexate tablets
  Interventions: Drug: 25 mg/week oral methotrexate tablets
- placebo (Placebo Comparator): 25 mg/week placebo tablets
  Interventions: Drug: 25mg/week oral placebo tablets

INTERVENTIONS:
Drug: 25 mg/week oral methotrexate tablets — active oral methotrexate drug
  Other Names: interventional drug
  Arms: methotrexate
Drug: 25mg/week oral placebo tablets — placebo comparator oral drug
  Arms: placebo

SUMMARY:
Osteoarthritis (OA) is a common disabling condition, for which no effective therapy currently exists. Synovitis has been demonstrated in hand OA imaging. Synovial inflammation due to the release of cytokines is an important cause of pain. Methotrexate (MTX) helps to decrease synovitis in many inflammatory joint diseases, particularly rheumatoid arthritis.

The aim of the present study is to assess the efficacy of MTX in decreasing pain and inflammation in symptomatic hand OA.

Methods: One hundred and twenty patients with American College of Rheumatology (ACR) clinical and radiographic criteria of primary knee OA with hand pain, [>4 on the 24-hour average pain severity scale (0-10) using mean of daily ratings from week preceding randomization] for > 14 days/month during 3 consecutive months preceding enrollment will be included in this randomized double-blind placebo-controlled trial. Patients meeting the eligibility criteria were randomized in a 1:1 ratio to receive either 25mg/week oral MTX (n=60) or placebo (n=60) together with their usual therapy provided the dosages were kept constant for 28 weeks. Pain will be assessed using the Visual Analogue pain Scale, (VAS, 0-100 mm). Functional assessment will be performed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Activities of daily living (ADL) scores. Alterations in dosage of analgesic/NSAID drugs used will be recorded. Safety and tolerability will also be assessed. Synovitis will be detected by ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* persistent pain
* synovitis

Exclusion Criteria:

* rheumatoid arthritis
* gout and pseudogout
* traumatic arthritis
* other secondary arthritis
* renal disease
* liver disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
pain reduction | 28 weeks
  The primary outcome will be pain reduction at 28 weeks compared to baseline using a Visual Analogue Pain Scale (VAS) 0-100 mm. Data will be collected at baseline and monthly up to 28 weeks to determine any change in results from those obtained at baseline.

SECONDARY OUTCOMES:
physical function improvement Functional assessment | 28 weeks
  Improvements in physical functioning McMaster Universities Osteoarthritis Index (WOMAC) subscores for pain, stiffness and function , the patient global assessment of the severity of knee OA measured on a 0-100 mm VAS. The physician-reported disease activity VAS was also recorded. Data will be collected at baseline and monthly up to 28 weeks to determine any change in results from those obtained at baseline.

OTHER OUTCOMES:
safety and tolerability | 28 weeks
  Safety and tolerability to treatment will be assessed at each visit. Safety will be assessed by identifying adverse events using open-ended questions and a checklist including common oral methotrexate side effects, physical examination and by laboratory assessment including complete blood picture and liver enzymes. Adverse events will be collected at each visit and up to 28 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt